CLINICAL TRIAL: NCT07262450
Title: Real-word Study to Assess Effectiveness of Seawater Nasal Sprays on Sinonasal Symptoms
Brief Title: Assessement of Effectiveness of Seawater Nasal Sprays on Sinonasal Symptoms
Acronym: SeaBridge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoire de la Mer (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A00394-45
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: URTI; Bronchiolitis; COVID - 19; Allergic Rhinitis; Chronic Rhinosinusitis (CRS); Post-surgery
MeSH Terms: conditions — Bronchiolitis; COVID-19; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Respimer® Hygiene-Prevention - Baby, kids, adults (Other): Respimer® Hygiene-Prevention - Baby, kids, adults - Lavage nasal Babies from 15 days, children & adults URTI; Bronchiolitis; Allergic rhinitis
  Interventions: Device: Respimer® Hygiene-Prevention -Baby, kids, adults
- Respimer® Hygiene-Prevention - Kids, adults (Other): Respimer® Hygiene-Prevention Kids, Adults -Nasal wash Children from 2 years & adults URTI; COVID-19; Allergic rhinitis; Chronic rhinosinusitis; Post-surgery
  Interventions: Device: Respimer® Hygiene-Prevention Kids, adults
- Respimer® Decongestion -Baby, kids, adults (Other): Respimer® Decongestion Baby, kids, adults - Nasal wash Babies from 2 months, children & adults URTI ; Allergic rhinitis; Chronic rhinosinusitis
  Interventions: Device: Respimer® Decongestion Baby, kids, adults
- Phytosun arôms® Hypertonic nasal wash - Children & adults (Other): Phytosun arôms® Hypertonic nasal wash Children from 6 years & adults URTI
  Interventions: Device: Phytosun arôms® Hypertonic nasal wash

INTERVENTIONS:
Device: Respimer® Hygiene-Prevention -Baby, kids, adults — 1-3 seconds spray in each nostril,
  * 4 to 6 times a day, in treatment of nasal symptoms.
  * 1 to 2 times a day, in hygiene and prevention
  Arms: Respimer® Hygiene-Prevention - Baby, kids, adults
Device: Respimer® Hygiene-Prevention Kids, adults — 1-2 seconds spray in each nostril,
  * 4 to 6 times a day, in treatment of nasal symptoms
  * 1 to 2 times a day, in hygiene and prevention
  Arms: Respimer® Hygiene-Prevention - Kids, adults
Device: Respimer® Decongestion Baby, kids, adults — Baby (2 months+): 1-3 seconds spray in each nostril, up to 3 times a day Children (2 y+) and adults: 1-3 seconds spray in each nostril, up to 6 times a day
  Arms: Respimer® Decongestion -Baby, kids, adults
Device: Phytosun arôms® Hypertonic nasal wash — 1 second spray in each nostril, 2-3 times a day.
  Arms: Phytosun arôms® Hypertonic nasal wash - Children & adults

SUMMARY:
The purpose of this post-market clinical investigation is to assess in a real-life setting, the effectiveness, usage, tolerance, safety and satisfaction of 4 isotonic and hypertonic seawater-based CE-marked nasal sprays.

The main questions it aims to answer are:

* Efficacy,
* Safety,
* Usage,
* Satisfaction, in real-life usage among infants, children, adults and pregnant or breastfeeding women suffering from acute and chronic sinonasal pathologies. The 4 medical devices under investigation will be used in accordance with their intended use, target populations and medical indications.

ELIGIBILITY:
Inclusion criteria:

* Subject's age and medical condition in compliance with the intended use and population
* Subjects who, from the investigator's judgement, should benefit from nasal wash in accordance with routine medical practice
* Subjects with at least two nasal symptoms of intensity ≥ 3 (6 modalities intensity SNOT-22 rating-scale) among the following:

  * Nasal blockage/nasal congestion/ stuffy nose;
  * Runny nose;
  * Need to blow/clear the nose;
  * Sneezing;
  * Thick nasal discharge/secretions;
  * Decreased sense of smell /taste (replaced by "noisy breathing/mouth breathing" for infants)
* Subjects with impaired nasal breathing (score ≥ 3, 6-modalities intensity rating-scale), induced by the presence of nasal symptoms
* For acute indications (only): subjects with symptoms started not later than 72 hours prior to enrolment (Day 0).
* For allergic rhinitis indication: perennial allergic rhinitis with and without seasonal allergic rhinitis
* For post-surgery indication: septoplasty and rhinoseptoplasty.
* Subject/parent willing to perform nasal wash following advices received from HCPs.
* Subjects (or parents for babies and children) agreeing to follow the study requirements during the whole study period (up to 3 months).
* Subject (or parent for baby and children) able to understand verbal and written local language and in capacity to fill-in questionnaire by himself.
* Subject having daily access to internet to answer online questionnaire.
* Subject or Parent/legal guardian of the subject has given freely and expressly her/his informed consent.
* Subject affiliated to the health social security system or beneficiary of an equivalent system

Non-inclusion criteria:

* Subject with contraindications according to each IFU.
* Hypersensitivity or known allergy to any component of the investigational products.
* Subject taking part in another clinical study or being in the exclusion period of another clinical study.
* Subject already using nasal wash to manage his nasal symptoms.
* Subject already included once in the study.
* Subject with a member of his household already included in the study if still in the follow-up phase.
* Subject deprived of liberty by administrative or judicial decision or under legal guardianship.

Min Age: 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1065 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Real-life effectiveness to improve nasal symptoms in case of acute and chronic sinonasal pathologies. | From Day 0 to Day 5 (acute indications: URTI, COVID-19, bronchiolitis) From Day 0 to Day 14 (chronic indications: allergic rhinitis, chronic rhinosinusitis, post-surgery)
  Change from baseline in nasal symptom intensity following initiation of nasal wash, based on the modified SNOT-22 rhinologic score. 6-modalities intensity Likert scale: 0=No problem; 1= Very mild problem; 2=Mild or slight problem; 3= Moderate problem; 4=Severe problem; 5=Problem as bad as it can be.

SECONDARY OUTCOMES:
Real-life effectiveness to reduce the intensity of individuals symptoms | From Day 0 to Day 14
  Daily change from baseline in individual symptoms intensity. 6-modalities intensity Likert scale.
Real-life effectiveness to reduce the intensity of additional extra nasal symptoms | From Day 0 to Day 14
  Daily change from baseline in additional extra nasal symptoms intensity. 6-modalities intensity Likert scale.
Real-life effectiveness to reduce the intensity of eyes symptoms | From Day 0 to Day 14
  Daily change from baseline in eyes symptoms intensity. Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ): 6-modalities scale.
Real-life effectiveness to reduce the daily intensity of symptoms | From Day 0 to Day 14
  Proportion of patients presenting a daily change in symptoms intensity; Modified SNOT-22: 6-modalities intensity Likert scale. Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ): 6-modalities scale
Real-life effectiveness to reduce the overall intensity of symptoms | From Day 0 to Day 14
  Daily change from baseline in the global modified SNOT-22 score and domains
Real-life effectiveness to reduce the frequency of sneezing | From Day 0 to Day 14
  Daily change from baseline in sneezing frequency. 5-modalities sneezing frequency scale
Real-life effectiveness to reduce the frequency of nose blowing | From Day 0 to Day 14
  Daily change from baseline in nose blowing frequency. 6-modalities nose blowing frequency scale
Real-life effectiveness to reduce the frequency of cough | From Day 0 to Day 14
  Daily change from baseline in cough frequency. 6-modalities Cough Symptom Score
Real-life effectiveness to relieve individual symptoms - Evolution | From Day 0 to Day 14
  Daily evolution of individual symptoms relief. Symptoms relief scale: 7-modalities scale
Real-life effectiveness to relieve individual symptoms | From Day 0 to Day 14
  Proportion of patients reporting a daily symptom relief. Symptoms relief scale: 7-modalities scale
Real-life effectiveness to relieve individual symptoms - 1st relief | From Day 0 to Day 14
  Number of days until first symptom relief. Symptoms relief scale: a 7-modalities scale
Real-life effectiveness to improve nasal breathing | From Day 0 to Day 14
  Daily change from baseline in nasal breathing difficulty. Nasal breathing difficulty scale: 6-modalities scale
Real-life effectiveness to improve nasal breathing - Onset | From Day 0 to Day 14
  Time to perceived improvement of nasal breathing. Nasal breathing scale: 7-modalities rating scale
Real-life effectiveness to improve nasal breathing - Duration | From Day 0 to Day 14
  Duration of improved nasal breathing. Improved nasal breathing scale: 7-modalities questionnaire
Real-life effectiveness to improve nasal breathing - Time interval | From Day 0 to Day 14
  Daily average time between two consecutive nasal washes. Open question whose unit of measurement is in hours
Real-life effectiveness to improve nasal blowing/removal of secretions | From Day 0 to Day 14
  Daily change from baseline in nose blowing/removal of secretions Easiness to blow the nose/remove secretions scale: 5-modalities rating scale
Real-life effectiveness to improve quality of secretions | From Day 0 to Day 14
  Daily change from baseline in quality of nasal secretions. Quality of nasal secretions scale: 4-modalities rating scale
Real-life effectiveness to improve quality of life | From Day 0 to Day 14
  Daily change from baseline in subjects' quality of life. QOL items of the modified SNOT-22 questionnaire: 6-modalities intensity Likert scale
Real-life effectiveness to improve quality of life - Energy | From Day 0 to Day 14
  Daily change from baseline in loss of energy. 4-modalities rating energy scale
Real-life effectiveness to improve quality of life - Daily activities | From Day 0 to Day 14
  Daily change from baseline in symptoms interference with daily activities. Symptom interference scale: 5-modalities rating scale
Real-life effectiveness to improve quality of life - Feeding difficulties | From Day 0 to Day 14
  Daily change from baseline in feeding difficulties. Babies's feeding difficulty scale: 0-10 VAS scale
Real-life effectiveness to improve quality of life - Baby and young child | From Day 0 to Day 14
  Daily change from baseline in cries frequency, irritability, comfort and wellbeing, overall behaviour.
  Baby and young child quality of life scale: 6-modalities rating scale.
Real-life effectiveness to improve quality of life of the family | From Day 0 to Day 14
  Daily change from baseline in family/parental quality of life. Family/parental quality of life scale: 6-modalities rating scale
Real-life effectiveness to limit nasal symptoms during winter and allergy seasons | From Day 15 to 3 months
  Number and proportion of subjects with nasal symptoms. Modified SNOT-22 self-questionnaire: 6-modalities intensity Likert scale
Real-life effectiveness to limit nasal symptoms during winter and allergy seasons. | From Day 15 to 3 months
  Number of nasal symptoms per subject. Modified SNOT-22 self-questionnaire: 6-modalities intensity Likert scale
Real-life effectiveness to limit nasal symptoms during winter and allergy seasons. | From Day 15 to 3 months
  Evolution of nasal symptoms intensity. SNOT-22 self-questionnaire: 6-modalities intensity Likert scale
Real-life effectiveness to limit nasal symptoms during winter and allergy seasons - Sneezing frequency. | From Day 15 to 3 months
  Evolution of sneezing frequency. 5-modalities sneezing frequency scale
Real-life effectiveness to limit nasal symptoms during winter and allergy seasons - Nose blowing. | From Day 15 to 3 months
  Evolution of nose blowing/Need to rub the nose frequency. 6-modalities nose blowing frequency scale
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons. | From Day 15 to 3 months
  Number and proportion of subjects with extra-nasal symptoms. Modified SNOT-22 self questionnaire: 6-modalities scale
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons. | From Day 15 to 3 months
  Number of extra-nasal symptoms per subject. Modified SNOT-22 self questionnaire: 6-modalities scale
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons. | From Day 15 to 3 months
  Evolution of extra-nasal symptoms intensity. Modified SNOT-22 self questionnaire: 6-modalities scale
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons - Eyes symptoms. | From Day 15 to 3 months
  Evolution of eyes symptoms intensity for allergic rhinitis sufferers. Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ):7-point Likert scale
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons. | From Day 15 to 3 months
  Evolution of modified SNOT-22 domains. Modified SNOT-22 self-questionnaire: 6-modalities scale
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons . | From Day 15 to 3 months
  Evolution of modified SNOT-22 global score. Modified SNOT-22 self-questionnaire: 6-modalities scale
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons - Cough, snoring, wake-up at night. | From Day 15 to 3 months
  Evolution of cough, snoring, wake up at night. Snoring, wake up at night (due to symptoms), cough frequency scale: 7-modalities rating scale
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons - Acute respiratory infections. | From Day 15 to 3 months
  Number and proportion of subjects with acute respiratory infection. Multiple-choice question regarding acute respiratory infection including the start date of the symptoms.
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons - Allergic rhinitis episodes. | From Day 15 to 3 months
  Number and proportion of subjects with acute allergic rhinitis episodes (for allergic rhinitis sufferers).
  Open question whose unit of measurement is in number of episodes.
Real-life effectiveness to limit extra-nasal symptoms during winter and allergy seasons - Asthma episodes. | From Day 15 to 3 months
  Number and proportion of subjects with asthma episodes/exacerbations (for allergic rhinitis sufferers).
  Open question whose unit measurement is in number of episodes.
Real-life effectiveness to improve nasal breathing quality during winter and allergy seasons. | From Day 15 to 3 months
  Evolution of nasal breathing score. Nasal breathing difficulty scale: 6-modalities scale
Real-life effectiveness to improve quality of life (QOL) during winter and allergy seasons. | From Day 15 to 3 months
  Evolution in modified SNOT-22 quality of life items. Modified SNOT-22 self-questionnaire: 6-modalities intensity Likert scale
Real-life effectiveness to improve quality of life (QOL) during winter and allergy seasons - Energy. | From Day 15 to 3 months
  Evolution in loss of energy. 4-modalities rating energy scale
Real-life effectiveness to improve quality of life (QOL) during winter and allergy seasons - Well-being & global health status | From Day 15 to 3 months
  Evolution of well-being and global health status. 0-10 VAS scale
Real-life effectiveness to improve quality of life (QOL) during winter and allergy seasons - Daily activities. | From Day 15 to 3 months
  Evolution of symptom interference with daily activities. 5-modalities rating scale
Real-life effectiveness to improve quality of life (QOL) during winter and allergy seasons - Practical problems. | From Day 15 to 3 months
  Evolution in practical problems (inconvenience of having to carry tissues/hankerchiefs, need to rub nose/eye, need to blow your nose repeatedly), for allergic rhinitis sufferers.
  6 modalities Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) scale.
Real-life effectiveness to limit the number of illness and missed days. | From Day 15 to 3 months
  Number of days with sickness / nasal symptoms. Open question whose unit of measurement is in number of days
Real-life effectiveness to limit the number of illness and missed days. | From Day 15 to 3 months
  Number and percentage of subjects with sickness days . Open question whose unit of measurement is in number of days
Real-life effectiveness to limit the number of illness and missed days. | From Day 15 to 3 months
  Number of missed days (work, school, daycare). Open question whose unit of measurement is in number of days
Real-life effectiveness to limit the number of illness and missed days. | From Day 15 to 3 months
  Number and percentage of subjects with missed days (work, school, daycare). Open question whose unit of measurement is in number of days
Real-life effectiveness to limit the impact on daily life for the family. | From Day 15 to 3 months
  Number of days of parental absence (work activities) due to baby/child's disease.
  Open question whose unit of measurement is in number of days
Real-life effectiveness to limit the impact on daily life for the family . | From Day 15 to 3 months
  Number and percentage of parents with missed days (work, activities). Open question whose unit of measurement is in number of days
Real-life effectiveness to limit the impact on daily life for the family. | From Day 15 to 3 months
  Number of days with impaired family/parental quality of life. Family/parental quality of life scale : 6-modalities rating scale
Real-life effectiveness to limit the impact on daily life for the family . | From Day 15 to 3 months
  Number and percentage of parents/family with impaired quality of life. Family/parental quality of life scale: 6 modalities rating scale
Real-life effectiveness to reduce the intake of concomitant medications during winter and allergy seasons. | From Day 15 to 3 months
  Number and percentage of subjects with intake of medications. Questions about name of the treatment, route of administration and number of days of use for each treatement
Real-life effectiveness to reduce the intake of concomitant medications during winter and allergy seasons. | From Day 15 to 3 months
  Number of days with intake of medications. Question about name of the treatment, route of administration and number of days of use for each treatement
Real-life effectiveness to reduce the intake of concomitant medications during winter and allergy seasons. | From Day 15 to 3 months
  Number and percentage of subjects in control group with re-introduction of nasal wash.
  Question about the name and format of the nasal wash product and number of days of use.
Real-life effectiveness to reduce the intake of concomitant medications during winter and allergy seasons. | From Day 15 to 3 months
  Evolution of allergic rhinitis treatment for allergic rhinitis sufferers. 3-modalities scale
Real-life effectiveness to reduce the evolution towards more severe form or complications. | From Day 15 to 3 months
  Number and percentage of subjects with severe symptoms intensity. Modified SNOT-22 self-questionnaire: 6-modalities intensity Likert scale
Real-life effectiveness to reduce the evolution towards more severe form or complications - Extra-nasal symptoms. | From Day 15 to 3 months
  Number and percentage of subjects with severe extra-nasal symptoms intensity. Modified SNOT-22 self-questionnaire: 6-modalities intensity Likert scale
Real-life effectiveness to reduce the evolution towards more severe form or complications - Eyes symptoms. | From Day 15 to 3 months
  Number and percentage of subjects with severe eyes symptom intensity. Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) scale: 7-point Likert scale
Real-life effectiveness to reduce the evolution towards more severe form or complications - Complications. | From Day 15 to 3 months
  Number and percentage of subjects with occurence of complications. Multiple-choice question.
Real-life effectiveness to reduce the evolution towards more severe form or complications - Asthma. | From Day 15 to 3 months
  Evolution of asthma symptoms frequency for asthma sufferers. 7-modalities frequency scale
Real-life effectiveness to reduce the evolution towards more severe form or complications - Asthma episodes. | From Day 15 to 3 months
  Number and percentage of subjects with asthma episodes/exacerbation for asthma sufferers.
  Open question
Real-life effectiveness to reduce the evolution towards more severe form or complications - Asthma intensity. | From Day 15 to 3 months
  Evolution of asthma symptoms intensity for asthma sufferers. 7-modalities scale
Real-life effectiveness to reduce the need for unplanned HCP care during winter and allergy seasons. | From Day 15 to 3 months
  Number and percentage of subjects consulting a HCP. Collection of unplanned HCP consultations because of nasal/respiratory symptoms
Real-life effectiveness to reduce the need for unplanned HCP care during winter and allergy seasons - Hospitalizations. | From Day 15 to 3 months
  Number and percentage of hospitalized subjects. Collection of hospitalizations due to nasal/respiratory symptoms
Real-life assessment of onset and duration of action and perceived effectiveness of the sprays - Onset. | From Day 15 to Month 3
  Time to perceived improvement of nasal breathing. 7 modalities rating scale.
Real-life assessment of onset and duration of action and perceived effectiveness of the sprays - Duration. | From Day 15 to Month 3
  Duration of improved nasal breathing. 7-modalities questionnaire
Real-life assessment of onset and duration of action and perceived effectiveness of the sprays. | From Day 15 to Month 3
  Daily average time between two consecutive nasal washes. Open question whose unit of measurement is in hours
Real-life assessment of onset and duration of action and perceived effectiveness of the sprays - Allergic rhinitis. | From Day 15 to Month 3
  Number and percentage of subjects with improved effectiveness of their usual allergic rhinitis treatment.
  7-modalities questionnaire
Real-life nasal sprays usage (posology, moment of use, usage versus medication) - Posology. | From Day 0 to Month 3
  Number of nasal wash per day and Number of days of use per week . 8-modalities posology questionnaire
Real-life nasal sprays usage (posology, moment of use, usage versus medication) - Moment of use. | From Day 0 to Month 3
  Moments of use of the nasal spray during the day. 7-modalities multiple choice question
Real-life nasal sprays usage (posology, moment of use, usage versus medication) - Co-usage with medications. | From Day 0 to Month 3
  Moments of use versus medications. Co-usage questionnaire.
Real-life nasal sprays usage (posology, moment of use, usage versus medication) - Occasion of use. | From Day 15 to Month 3
  Occasion of use during the prevention phase. Multiple-choice question
Real-life nasal sprays usage (posology, moment of use, usage versus medication) - Baby nasal aspirator. | From Day 0 to Month 3
  Complementary usage of a baby nasal aspirator. 7-modalities frequency scale
Real-life nasal sprays usage (posology, moment of use, usage versus medication) - Child autonomy. | From Day 0 to Month 3
  Child's autonomy in using the nasal spray. Multiple-choice question
Real-life assessment of satisfaction and willingness to reuse and recommandation of the nasal sprays - Satisfaction. | From Day 0 to Month 3
  Number and percentage of subjects satisfied with the use of the nasal spray. 5-modalities satisfaction scale.
Real-life assessment of satisfaction and willingness to reuse and recommandation of the nasal sprays - Perceived sensation. | From Day 0 to Month 3
  Perceived sensation after application. 5-modalities sensory scale.
Real-life assessment of satisfaction and willingness to reuse and recommandation of the nasal sprays - Perceived effectiveness. | From Day 0 to Month 3
  Global perceived effectiveness of the nasal spray. 6-modalities rating scale
Real-life assessment of satisfaction and willingness to reuse and recommandation of the nasal sprays - Practicality. | From Day 0 to Month 3
  Practicality of the product, easiness to use. 6-modalities technical performance agreement scale.
Real-life assessment of satisfaction and willingness to reuse and recommendation of the nasal sprays - Reuse and recommend. | From Day 0 to Month 3
  Number and percentage of subjects with willingness to reuse, willingness to recommend the nasal spray.
  4-modalities scale
Real-life assessment of satisfaction and willingness to reuse and recommandation of the nasal sprays - Educational content. | From Day 0 to Month 3
  Usefulness of the educational content (tutorial and tips). Multiple choice satisfaction questionnaire.
Assessment of the safety and tolerance of the nasal sprays - Tolerance. | From Day 0 to Month 3
  Evolution of tolerance to the nasal spray. 4-modalities scale.
Assessment of the safety and tolerance of the nasal sprays - Safety. | From Day 0 to Month 3
  Number and percentage of incidents reported during the clinical investigation. Number and percentage of subjects reporting incidents during the clinical investigation.
  Collection of incidents and adverse events (nature, dates of occurrence and evolution).

CONTACTS AND LOCATIONS:
Locations (32):
- France (32):
  - CHU Bordeaux, Bordeaux
  - Pharmacie de la Faïncerie, Bourg-la-Reine
  - Pharmacie Marine, Cabourg
  - Pharmacie Daguet, Châteauroux
  - Pharmacie des verts coteaux, Châtenay-Malabry
  - Pharmacie Lombard, Châtenay-Malabry
  - Maison Médicale Avicenne, Chevaigné
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Kap Santé, Courrières
  - Pharmacie de la Liberté, Falaise
  - Maison médicale Heyrieux, Heyrieux
  - CHD Vendée, La Roche-sur-Yon
  - CKRF Marcq en Baroeul, Marcq-en-Barœul
  - Centre de Kinésithérapie spécialisé en rééducation respiratoire - Marseille, Marseille
  - La Maison du Souffle, Metz
  - Centre médical Chamberte, Montpellier
  - CHU Poitiers, Poitiers
  - Pharmacie du Pot d'Etain, Pont-Audemer
  - Pharmacie DRAPEAU, Pont-Saint-Martin
  - Cabinet de kinésithérapie respiratoire Sophie Jacques, Rennes
  - Pharmacie Deroche, Roézé-sur-Sarthe
  - Pharmacie Girard, Saint-Colomban
  - Clinique Saint-Jean, Saint-Jean-de-Védas
  - Centre de santé respiratoire Saint Paul Lès Dax, Saint-Paul-lès-Dax
  - Pharmacie des Corsaires, St-Malo
  - Pôle Santé de Réadaptation Toulouse Ouest, Toulouse
  - CRKF Tourcoing, Tourcoing
  - Maison médicale Belencontre, Tourcoing
  - Maison médicale de la Bourgogne, Tourcoing
  - Centre respiratoire de Valenciennes, Valenciennes
  - Cabinet de Kinésithérapie HODOROABA Vincent, Wissous
  - Pharmacie St-Exupery, Wissous

IPD SHARING:
Plan to Share IPD: No